CLINICAL TRIAL: NCT01710748
Title: Reservoir-Based Polymer-Free Amphilimus-Eluting Stent Versus Polymer-Based Everolimus-Eluting Stent in Diabetic Patients (RESERVOIR) Trial
Brief Title: Reservoir-Based Polymer-Free Amphilimus-Eluting Stent Versus Polymer-Based Everolimus-Eluting Stent in Diabetic Patients
Acronym: RESERVOIR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Spanish Society of Cardiology (Other)
Responsible Party: Principal Investigator, Dr Rafael Romaguera, Dr. Rafael Romaguera, Spanish Society of Cardiology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SEC-RES-2012-01
Record Dates: First submitted 2012-10-17; First posted 2012-10-19 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Coronary Artery Disease; Diabetes Mellitus
Keywords: Percutaneous coronary intervention; Drug eluting stent; Neointimal hyperplasia; Diabetes Mellitus
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polymer-Based Everolimus-Eluting Stent (Active Comparator): Polymer-Based Everolimus-Eluting Stent
  Interventions: Device: Polymer-Based Everolimus-Eluting Stent
- Polymer-Free Amphilimus-Eluting Stent (Experimental): Reservoir-Based Polymer-Free Amphilimus-Eluting Stent
  Interventions: Device: Polymer-Free Amphilimus-Eluting Stent

INTERVENTIONS:
Device: Polymer-Based Everolimus-Eluting Stent — Polymer-Based Everolimus-Eluting Stent
  Other Names: Xience Coronary Stent System
  Arms: Polymer-Based Everolimus-Eluting Stent
Device: Polymer-Free Amphilimus-Eluting Stent — Reservoir-Based Polymer-Free Amphilimus-Eluting Stent
  Other Names: Cre8 Coronary Stent System
  Arms: Polymer-Free Amphilimus-Eluting Stent

SUMMARY:
This study is a prospective, randomized controlled, single blind, two-arm, multicenter clinical evaluation.

Diabetic patients (n=112) with de novo coronary artery disease will be randomized to one of the 2 treatment arms: 1) Reservoir-Based Polymer-Free Amphilimus-Eluting Stent or 2) Polymer-Based Everolimus-Eluting Stent.

The purpose of this study is to determine whether Polymer-Free Amphilimus-Eluting Stent implantation is effective in reducing neointimal hyperplasia as compared to Polymer-Based Everolimus-Eluting Stent in diabetic patients, using Optical Coherence Tomography (OCT) as the primary imaging modality.

DETAILED DESCRIPTION:
In patients with diabetes mellitus (DM), drug eluting stents (DES) have been shown to be associated with greater neointimal suppression than bare-metal stents. However, there is an ongoing debate on the optimal drug-eluting stent in diabetic patients.

This study is a prospective, randomized controlled, single blind, two-arm, multicenter clinical evaluation.

Diabetic patients (n=112) with de novo coronary artery disease will be randomized to one of the 2 treatment arms: 1) Reservoir-Based Polymer-Free Amphilimus-Eluting Stent or 2) Polymer-Based Everolimus-Eluting Stent.

The purpose of this study is to determine whether Polymer-Free Amphilimus-Eluting Stent implantation is effective in reducing neointimal hyperplasia as compared to Polymer-Based Everolimus-Eluting Stent in diabetic patients, using Optical Coherence Tomography (OCT) as the primary imaging modality.

ELIGIBILITY:
Clinical Inclusion Criteria:

* Subject is eligible for PCI.
* Subject has symptomatic coronary artery disease (stable/unstable angina or Non-ST elevation myocardial infarction).
* Subject has known DM.

Angiographic Inclusion Criteria:

* Presence of 1 or 2 de novo native coronary artery lesions (maximum 1 lesion per epicardial coronary artery), with a visual estimation stenosis ≥ 50%.
* Target lesion length 12-25mm, reference diameter 2.5-3.5mm.

Clinical Exclusion Criteria:

* ST-segment elevation myocardial infarction <48h
* Presence of cardiogenic shock pre-procedure
* Contra-indications to dual antiplatelet therapy for 12 months
* Left Ventricular Ejection Fraction ≤30%
* GFR<30 ml/min/m2
* Target vessel has been treated previously
* Platelet count <75000/mm3 or >700000/mm3
* Immunosuppressive therapy
* Has received or waiting list for any transplant
* Life-threatening disease with a life expectancy of < 12 months
* Pregnant or breast feeding patient
* Inability to provide informed consent

Angiographic Exclusion Criteria:

* TIMI flow ≤ 1 prior to guide wire crossing
* There is an additional lesion within the target vessel planned to be treated within the next 12 months
* Target vessel is a saphenous vein graft
* Target vessel is the left main, ostial LAD and/or ostial LCX.
* Prior PCI of the target lesion (restenosis)
* Lesion cannot be covered by a single stent (unplanned bailout stenting is allowed)
* Involved side branch ≥2.5mm by visual estimation
* Rotablator, ELCA or brachytherapy
* Severe calcification of target lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-07 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Neointimal hyperplasia volume obstruction | 9 months
  The primary endpoint is assessed by Optical Coherence Tomography. It is defined as neointimal hyperplasia volume (mm3) divided by the stent volume multiplied by 100.

SECONDARY OUTCOMES:
Percentage of uncovered struts | 9 months
  This endpoint is assessed by Optical Coherence Tomography. Struts are classified as uncovered if any part of the strut is visibly exposed to the lumen, or covered if a layer of tissue is visible over all the reflecting surfaces.
Percentage of malapposed struts | 9 months
  This endpoint is assessed by Optical Coherence Tomography. Apposition is assessed strut by strut by measuring the distance between the strut marker and the lumen contour. Struts with distance to lumen contour larger than the sum of strut + polymer thickness are considered malapposed. This results in incomplete strut apposition thresholds of 89 µm for the Xience Prime and 80 µm for the Cre8 stent. Struts located at the ostium of side branches, with no vessel wall behind, are excluded from the analysis of apposition.
Maximum percentage of NIH cross-sectional obstruction | 9 months
  This endpoint is assessed by Optical Coherence Tomography. Percentage of NIH cross-sectional obstruction is defined as the NIH area (mm2) divided by the stent area multiplied by 100.
Cardiac death | 12 months
  Death related to cardiac causes; if the cause of death cannot be determined, it will be also categorized as cardiac.
Probable or definite stent thrombosis | 12 months
  Stent thrombosis is considered according to the Academic Research Consortium definitions
Target vessel failure | 12 months
  Target vessel failure is defined as a composite endpoint of cardiac death, target vessel myocardial infarction and clinically indicated revascularization of the target vessel.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Romaguera, MD, Principal Investigator — Spanish Society of Cardiology
Locations (4):
- Spain (4):
  - Hospital Clínic i Provincial, Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona, Barcelona
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Virgen de la Arrixaca, Murcia, Murcia

REFERENCES:
- [Derived] Romaguera R, Gomez-Hospital JA, Gomez-Lara J, Brugaletta S, Pinar E, Jimenez-Quevedo P, Gracida M, Roura G, Ferreiro JL, Teruel L, Montanya E, Fernandez-Ortiz A, Alfonso F, Valgimigli M, Sabate M, Cequier A. A Randomized Comparison of Reservoir-Based Polymer-Free Amphilimus-Eluting Stents Versus Everolimus-Eluting Stents With Durable Polymer in Patients With Diabetes Mellitus: The RESERVOIR Clinical Trial. JACC Cardiovasc Interv. 2016 Jan 11;9(1):42-50. doi: 10.1016/j.jcin.2015.09.020. PMID 26762910
- [Derived] Romaguera R, Brugaletta S, Gomez-Lara J, Pinar E, Jimenez-Quevedo P, Gracida M, Roura G, Ferreiro JL, Teruel L, Gomez-Hospital JA, Montanya E, Alfonso F, Valgimigli M, Sabate M, Cequier A. Rationale and study design of the RESERVOIR trial: a randomized trial comparing reservoir-based polymer-free amphilimus-eluting stents versus everolimus-eluting stents with durable polymer in patients with diabetes mellitus. Catheter Cardiovasc Interv. 2015 Mar;85(4):E116-22. doi: 10.1002/ccd.25728. Epub 2014 Nov 27. PMID 25380051